CLINICAL TRIAL: NCT05256407
Title: Digital Support for Parents of Children in Child Health Care - an Evaluation of an Intervention in Primary Health Care
Brief Title: Digital Support for Parents of Children in Child Health Care
Acronym: LValan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: Västernorrland County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Asa Hornsten, Professor, Umeå University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UmU-2021-LValan
Record Dates: First submitted 2021-09-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Parenting; Children, Only; Health Care Seeking Behavior; Health Knowledge, Attitudes, Practice; Nurse-Patient Relations
MeSH Terms: conditions — Patient Acceptance of Health Care; Behavior | interventions — Methods

STUDY DESIGN:
Intervention Model Description: prospective case/control intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, digital support (Experimental): Parents are offered participation in a digital channel consisting of video consultations, parental support gruops and parental education.
  Interventions: Other: Intervention, digital support
- Control, usual care (No Intervention): Usual child health care.

INTERVENTIONS:
Other: Intervention, digital support — Internet based support of parents in child health care. Various options and choices includes parental education, digital meetings with child health nurse and peer groups
  Arms: Intervention, digital support

SUMMARY:
Becoming a parent is a life-changing event that can be both gratifying and stressful. As a parent, one is responsible for another person, where there sometimes is a need for new information, knowledge, and advice to live up to the new requirements that a changing family situation requires. The objective of this study is to develop and evaluate a new digital channel in child health care for support of parents in child health care issues with particular focus on eHealth literacy and satisfaction with care. An intervention is planned to run over eight months and will be evaluated in an intervention- and control group (from another health care centre) at baseline, 4 months and at 8 months follow-up. Data includes interviews and questionnaires about parental stress and eHealth literacy as well as satisfaction with care. Data will be analysed with qualitative and statistical methods. Expected outcomes is reduced parental stress and increased satisfaction with child health care.

ELIGIBILITY:
Inclusion Criteria:

* Swedish speaking parents with children (0-6 years) in Swedish child health care

Exclusion Criteria:

* Parents who are registered at an address other than their child
* Parents younger than 16 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Parental Stress Scale | Parental stress at baseline
  The scale consists of 17 questions graded from 1 to 5, where 1 indicates "Do not agree at all" and 5 is "Agree completely". A total is calculated by adding all items together to obtain a score ranging from 18 to 90, with higher scores indicating higher levels of parental stress.
Parental Stress Scale | Change Parental stress at 4 months
  The scale consists of 17 questions graded from 1 to 5, where 1 indicates "Do not agree at all" and 5 is "Agree completely". A total is calculated by adding all items together to obtain a score ranging from 18 to 90, with higher scores indicating higher levels of parental stress.
Parental Stress Scale | Change Parental stress at 8 months
  The scale consists of 17 questions graded from 1 to 5, where 1 indicates "Do not agree at all" and 5 is "Agree completely". A total is calculated by adding all items together to obtain a score ranging from 18 to 90, with higher scores indicating higher levels of parental stress.

SECONDARY OUTCOMES:
eHealth Scale | eHealth literacy at baseline
  The eHeals scale consists of 10 questions in five ratings where 1 is "do not agree at all" and 5 "fully agree". Total scores of the eHEALS are summed to range from 8 to 40, with higher scores representing higher self-perceived eHealth literacy.
eHealth Scale | Increased eHealth literacy at 4 months
  The eHeals scale consists of 10 questions in five ratings where 1 is "do not agree at all" and 5 "fully agree". Total scores of the eHEALS are summed to range from 8 to 40, with higher scores representing higher self-perceived eHealth literacy.
eHealth Scale | Increased eHealth literacy at 8 months
  The eHeals scale consists of 10 questions in five ratings where 1 is "do not agree at all" and 5 "fully agree". Total scores of the eHEALS are summed to range from 8 to 40, with higher scores representing higher self-perceived eHealth literacy.

OTHER OUTCOMES:
VAS Scale | Satisfaction with child health care at baseline
  The VAS scale consists of a line with a cross marker where participants can make crosses according to a 5 degree scale in 3 different questions. The line is divided into 5 points with 1 cm distance where marking 1 from the left is graded "not at all" to the last on the right side of the line is 5 "Completely". Total scores of the VAS are summed to range from 3 to 15, with higher scores representing higher levels of degrees.
VAS Scale | Satisfaction with child health care at 4 months
  The VAS scale consists of a line with a cross marker where participants can make crosses according to a 5 degree scale. The line is divided into 5 points with 1 cm distance where marking 1 from the left is graded "not at all" to the last on the right side of the line is "Completely". Total scores of the VAS are summed to range from 3 to 15, with higher scores representing higher levels of degrees.
VAS Scale | Satisfaction with child health care at 8 months
  The VAS scale consists of a line with a cross marker where participants can make crosses according to a 5 degree scale. The line is divided into 5 points with 1 cm distance where marking 1 from the left is graded "not at all" to the last on the right side of the line is "Completely". Total scores of the VAS are summed to range from 3 to 15, with higher scores representing higher levels of degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Västernorrland, Örnsköldsvik, Sweden

IPD SHARING:
Plan to Share IPD: No